CLINICAL TRIAL: NCT01964209
Title: Initial Validation of the Vanderbilt Attention Deficit Hyperactive Disoder (ADHD) Measure for Adolescent Patients in the Integrated Clinical Information Sharing System (ICISS) Project
Brief Title: Initial Validation of the Vanderbilt ADHD Measure for Adolescent Patients in the ICISS Project
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Joshua Borus, Staff Physician, Boston Children's Hospital
Other Study IDs: 83064
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: ADHD
Keywords: ADHD; Validation; Quality Improvement; Vanderbilt; Conners 3rd Edition; ADHD Measures; ADHD Adolescent; ADHD Questionnaire; ICISS; Integrated Clinical Information Sharing System
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: This is a psychometric study of a screening tool for ADHD, so we will not be administering any treatments or interventions.

SUMMARY:
This proposal is to evaluate the reliability and validity of the Vanderbilt ADHD screening tool for use with adolescents and young adults aged 13-21 years. The Vanderbilt is a previously developed, freely available set of parent- and teacher-report questionnaires designed to identify ADHD and related disorders in children. The Vanderbilt measures have been chosen for inclusion in the new computerized Integrated Clinical Information Sharing System (ICISS) being rolled out in five Boston Children's Hospital (BCH) departments/divisions (Adolescent/Young Adult Practice, Children's Hospital Primary Care Center, Developmental Medicine Center, Department of Neurology, Department of Psychiatry). The Vanderbilt was developed and validated for use among children up to age 12 years (Wolraich et al., 2003; Wolraich et al., 2013; Bard et al., 2013), and little is known about its appropriateness for use among older youth. In addition, there is no self-report version of the Vanderbilt that can be administered directly to adolescents and young adults (ages 13-21 years), for whom parents and teachers are often less knowledgeable reporters. To address these shortcomings, a multidisciplinary team of BCH adolescent health clinicians and researchers modified the parent and teacher Vanderbilt questionnaires to make them age-appropriate for adolescents and young adults and created a complementary self-report version for adolescents and young adults. The goal of the current study is to 1) assess the feasibility and acceptability of online administration through the ICISS system of the new parent, teacher, and youth self-report Vanderbilt measures among adolescent and young adult BCH patients aged 13-21 years; 2) test their reliability in terms of internal consistency reliability, temporal stability of responses over a one-month test-retest, and inter-rater agreement across all informants (parents, teachers, and youths); and 3) test their validity by evaluating their convergence with a similar set of ADHD screening tools, the Conners scales, already validated for use with adolescents and young adults.

DETAILED DESCRIPTION:
Background and Specific Aims:

Study Design: We will use the ICISS system's capacity for prospective and ongoing collection of data from enrolled patients and their families to conduct our prospective, longitudinal study consisting of a baseline assessment at enrollment into ICISS, a one-month re-test assessment, and a follow-up assessment at either 3 months for patients who were newly-diagnosed with ADHD or had a change in medication, or 6 months for patients with an established diagnosis and no medication changes.

Recruitment and Consent: Once a patient has enrolled in ICISS, they will be asked if they wish to participate in the modified Vanderbilt validation study, initially by phone call. Some patients and/or their parents will want to discuss this in person or may not be reached by phone call, in which case the research assistant will meet with them at the clinic visit. This will take place in a quiet, confidential space.

However, with adolescents it is typical that the parent is not present at the clinic visit. The Vanderbilt validation study will then be discussed with the parent verbally by phone and consent will be implicit in answering the two Conners questionnaires when sent online. Interested and eligible patients will be reminded in this email that participation in this research study is completely voluntary, that a decision not to participate will not affect their medical care in any way and that they may withdraw from the study at any time.

As participation in this study consists simply of answering two Conners questionnaires which represent the standard of care for ADHD both nationally and in our clinics, presents virtually no risk to the participant above the minimal risks associated with the general ICISS study, and the parent, participant and teacher all have the option to simply not respond to the email requesting Conners completion for this study.

Data Collection and Measures: The increase in effort to collect the additional data needed for our study will be small as most of these measures are already being collected as part of the larger ICISS implementation. The added time for each participant to complete the Conners measures is marginal, on the order of 30 minutes total over a few interactions. After enrollment into ICISS, all eligible patients aged 13-21 years will be asked to complete the baseline youth self-report Vanderbilt-Long Form questionnaire and their parents the Parent version. In addition, patients 13-18 years will have teachers complete the Teacher version. All Long-Form versions include 18 items assessing the frequency (using a response scale of 0=Never, 1=Occasionally, 2=Often, 3=Very often) of symptoms and behaviors indicative of the predominant subtype of ADHD (Inattentive, Hyperactive/Impulsive, or Combined). Additionally, all three versions screen for Anxiety/Depression (7 items) and Oppositional-Defiant Disorder (8 items), disorders that often co-occur with ADHD. Lastly, only the Parent and Teacher versions include items assessing Conduct Disorder and School Performance (e.g., academic performance, peer relations, classroom behavior, and assignment completion). To assess test-retest reliability, we will again administer the Long-Forms at one-month follow-up. However, for subsequent follow-ups (i.e., 3- or 6-months), we will administer the Short-Form for all three Vanderbilt measures, which is the Long-Form but with the omission of Anxiety/Depression and Oppositional-Defiant disorder items. We will also collect the following data to address each of our study aims:

Aim 1: Feasibility and Acceptability: We will record patient, parent, and teacher response and completion rates for each Vanderbilt administration. We will also measure the length of time it takes for them to complete the Long Form (administered at baseline and one-month follow-up) and Short Form (administered monthly thereafter), and provide comment fields so that they can describe any difficulties they may have had in answering any of the questions.

Aim 2: Test-Retest and Inter-Rater Reliability: All patients, parents, and teachers will again receive their respective Long-Form version of the Vanderbilt at one-month follow-up. As part of the ICISS system, they will receive an email prompting them to complete the forms and submit them electronically to ICISS where they will be made available to the team and the patient's clinician. We will examine test-retest only for those patients who had no new medications or changes in their medications and stable symptoms during the intervening month. We will use the following two items to identify these patients: 1) "Since your/your child's last medical appointment in the Adolescent Practice, have there been any changes in your/his/her ADHD-related medications or therapies?" (Yes, No, I/My child do/does not receive ADHD-related medications or therapies); and 2) "In general, how would you describe your/your child's ADHD symptoms since your/his/her last medical appointment in the Adolescent Practice?" (They have improved, They have stayed about the same, They have gotten worse). We will only include patients for whom both the parent and patient reports indicate no changes in symptoms or medications/therapies. We will examine both item-level retest agreement as well as reliability of the overall screening outcome within each Vanderbilt domain (e.g., whether criteria are met for ADHD [and the predominant subtype], Oppositional-Defiant Disorder, Anxiety/Depression, etc.).

We will also examine, when data are available, the level of "inter-rater" agreement, at the domain level, across screening results obtained from youth, parent, and teacher forms.

Aim 3: Concurrent and Known-Groups Validity: For patients ages 13-18 years, we will administer concurrent with the Vanderbilt at all assessment time points (see Study Design), the Conners 3rd Edition Self Report Scale - Short Form (39 items); the Parent Rating Scale (43 items); and the Teacher Rating Scale (39 items). For patients ages 19-21 yrs, we will administer the Conners Adult ADHD Rating Scale Self-Report - Screening Version (30 items), and ask parents to complete the corresponding Observer Report - Screening Version (30 items) (Erhardt et al, 1999; Van Voorhees et al., 2011). We opted to use the adult ADHD rating scales for patients aged 19 years or older since the Conners 3rd Edition measures have only been validated up to age 18 years. We also opted to drop the teacher-based assessment for patients older than 18 years due to concern that many teachers would be unable to assess participants given minimal personal interaction in most college classes and the participant's possible desire to keep ADHD diagnosis private. To test the ability of the Vanderbilt scores to differentiate adolescents who are expected to differ (known-groups validity), we will administer 1) a modified version of the Clinical Global Impression Scale [CGIS], a single-item measure of adolescent global functioning (Busner & Targum, 2007) that parents and youth both complete; 2) among patients 13-18 years, the PedsQL-Family Impact Module (Varni et al., 2004) a 36-item parent-report measure of the impact a child's health condition is having on parent/family quality of life; and among patients 19-21 years, the 29-item Adult ADHD Quality of Life Questionnaire (AAQoL) (Matza et al., 2007). We will use these quality of life and functioning measures to categorize youth into low, medium, and high symptom-severity groups, and assess the ability of the Vanderbilt measures to discriminate these groups. Finally, we will identify those patients who experience a change in their scores on the validation measures (Conners, CGIS, PedsQL-Family Impact Module) over the follow-up period (3 months for newly-diagnosed or medication-change patients, 6 months for established/no-medication-change patients) and assess the Vanderbilt's ability to detect that change.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 13-21 who already have an ADHD diagnosis or are being evaluated for ADHD.
* Parent/guardian will be asked to participate for patients ages 13-21.
* Teachers will be asked to participate for patients ages 13-21.
* All informants should be able to read and understand English at a 5th grade reading level; and enrolled in the ICISS system.

Exclusion Criteria:

* Cognitive impairment or developmental delay.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Boston Children's Hospital patients which will be recruited from the following divisions: Adolescent/Young Adult Practice, Developmental Medicine Center and Department of Psychiatry.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2018-07 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Reliability of the Vanderbilt | One month after initial administration of Vanderbilt
  We will assess for each measure the level of internal consistency reliability, temporal stability of responses over a one-month test-retest, and inter-rater agreement across all informants (parents, teachers, and youths).

SECONDARY OUTCOMES:
Validity of Vanderbilt | One month after initial administration of Conners
  We will assess construct validity by evaluating the degree to which the Vanderbilt measures show convergence with a similar set of ADHD screening tools, the Conners scales, already validated for use with adolescents up to age 18 years (the Conners 3rd Edition Parent, Teacher, and youth Self-Report scales) and with young adults ages 19-21 years (the Conners Adult ADHD Rating Scale - Self-Report and Observer-Report versions).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Borus, MD,MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Adolescent/ Young Adult Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barbaresi WJ, Katusic SK, Colligan RC, Pankratz VS, Weaver AL, Weber KJ, Mrazek DA, Jacobsen SJ. How common is attention-deficit/hyperactivity disorder? Incidence in a population-based birth cohort in Rochester, Minn. Arch Pediatr Adolesc Med. 2002 Mar;156(3):217-24. doi: 10.1001/archpedi.156.3.217. PMID 11876664
- [Background] Bard DE, Wolraich ML, Neas B, Doffing M, Beck L. The psychometric properties of the Vanderbilt attention-deficit hyperactivity disorder diagnostic parent rating scale in a community population. J Dev Behav Pediatr. 2013 Feb;34(2):72-82. doi: 10.1097/DBP.0b013e31827a3a22. PMID 23363972
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Conners CK, Wells KC, Parker JD, Sitarenios G, Diamond JM, Powell JW. A new self-report scale for assessment of adolescent psychopathology: factor structure, reliability, validity, and diagnostic sensitivity. J Abnorm Child Psychol. 1997 Dec;25(6):487-97. doi: 10.1023/a:1022637815797. PMID 9468109
- [Background] Erhardt, D., Epstein, J. N., Conners, C. K., Parker, J. D., Sitarenios, G. (1999, October). Self-ratings of ADHD symptoms in adults II: reliability, validity, and diagnostic sensitivity. Journal of Attention Disorders, 3 (3), 153-158
- [Background] Klassen AF, Miller A, Fine S. Health-related quality of life in children and adolescents who have a diagnosis of attention-deficit/hyperactivity disorder. Pediatrics. 2004 Nov;114(5):e541-7. doi: 10.1542/peds.2004-0844. PMID 15520087
- [Background] Matza LS, Johnston JA, Faries DE, Malley KG, Brod M. Responsiveness of the Adult Attention-Deficit/Hyperactivity Disorder Quality of Life Scale (AAQoL). Qual Life Res. 2007 Nov;16(9):1511-20. doi: 10.1007/s11136-007-9254-9. Epub 2007 Sep 12. PMID 17874207
- [Background] Van Voorhees EE, Hardy KK, Kollins SH. Reliability and validity of self- and other-ratings of symptoms of ADHD in adults. J Atten Disord. 2011 Apr;15(3):224-34. doi: 10.1177/1087054709356163. Epub 2010 Apr 27. PMID 20424007
- [Background] Varni JW, Limbers CA, Burwinkle TM. Parent proxy-report of their children's health-related quality of life: an analysis of 13,878 parents' reliability and validity across age subgroups using the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jan 3;5:2. doi: 10.1186/1477-7525-5-2. PMID 17201923
- [Background] Wolraich ML, Bard DE, Neas B, Doffing M, Beck L. The psychometric properties of the Vanderbilt attention-deficit hyperactivity disorder diagnostic teacher rating scale in a community population. J Dev Behav Pediatr. 2013 Feb;34(2):83-93. doi: 10.1097/DBP.0b013e31827d55c3. PMID 23363973
- [Background] Wolraich ML, Lambert W, Doffing MA, Bickman L, Simmons T, Worley K. Psychometric properties of the Vanderbilt ADHD diagnostic parent rating scale in a referred population. J Pediatr Psychol. 2003 Dec;28(8):559-67. doi: 10.1093/jpepsy/jsg046. PMID 14602846